CLINICAL TRIAL: NCT05208606
Title: Advancing Palliative Care in Northern Plains American Indians: Living Well With Serious Illness "Wicokuje Sica Tuha Akisniya Wiconi" - Wawokiya Health Advocate Intervention
Brief Title: Living Well With Serious Illness "Wicokuje Sica Tuha Akisniya Wiconi": Wawokiya Health Advocate Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: South Dakota State University (Other); Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Principal Investigator, Katrina Armstrong, M.D., Physician-In-Chief, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021P003376
Record Dates: First submitted 2021-12-28; First posted 2022-01-26 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2023-07

CONDITIONS: Cancer
Keywords: American Indians; Community Health Worker; Palliative Care; Native American; Navigation; Lay Health Worker; Cancer Navigation
MeSH Terms: conditions — Neoplasms | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: A novel model will be used in alignment with community feedback on study design. Patients will be allocated to the intervention arm as dictated by interventionist panel capacity. Patients will be added to a waitlist "control" arm as dictated by intervention arm capacity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wawokiya Health Advocate (Experimental): Patients and caregivers allocated to the Wawokiya Health Advocate arm will receive a palliative intervention consisting of regular needs assessments and home visits. After the first 2 visits, visits will occur bi-weekly, though a WHA may increase or decrease frequency of visits pending patient and caregiver needs and cancer status. The first two study visits will follow the same broad structure-structure of follow up visits will be flexible based on patient and caregiver needs. The location of study visits will vary and may include the local IHS site, cancer centers, and the patient's home depending on health status. Patients will be randomized to either receive home visits upon enrollment or be placed on a waitlist.
  Interventions: Behavioral: Wawokiya Health Advocate
- Waitlist Arm (No Intervention): Patients enrolled into the waitlist group will not receive any additional services beyond what is available to them in their standard course of care. Patients randomized to the waitlist group will be asked to identify a primary caregiver upon enrollment. Data collection procedures will occur as described below. While on the waitlist, any services available for patients and their families will be according to the standards of their local providers and primary cancer providers.

INTERVENTIONS:
Behavioral: Wawokiya Health Advocate — Study visits 1 and 2 will follow the same broad procedures. Subsequent visits will be structured around needs. WHAs will cover multiple domains of assessment utilizing a visit guide.
  Visit 1: Specific topics covered in this visit will include; 1) an explanation of palliative care, study, and WHA role and 2) mapping of providers/family/caregivers The WHA will arrange dates and times for future visits.
  Visit 2: Occurs 1 week after the first visit. WHAs will begin to assess patient needs utilizing a needs assessment tool. Specific topics covered will include: 1) Documentation of disease history 2) Needs assessment screen
  Following Visits: After visit 2, activities will be based on needs assessed. Activities may entail: 1) Review of palliative care and WHA role, 2) Assessment of needs, 3) Addressing needs 3) Exploring goals of care.
  We anticipate patients will receive an average of 2-3 WHA visits per month. Investigators will hold regular supervisory meetings with the WHA.
  Other Names: Community Health Worker
  Arms: Wawokiya Health Advocate

SUMMARY:
Informed by a Community Advisory Board (CAB) and community assessments performed in the first phase of work funded through R01CA240080, this study will test a wawokiya (one who helps) health advocate (WHA)-based palliative care intervention that aims to improve the wellbeing of patients with cancer. In alignment with community guidance, patients will be allocated to an intervention arm or a waitlist arm as dictated by capacity. For those patients receiving the intervention, palliative care trained WHAs will perform regular home visits to assess the needs of patients seriously ill with cancer (as defined by a referring provider) and their caregivers, and work to address those needs using their training and identified community resources. The frequency of visits / calls will be determined based on level of need. The specific aims are listed below.

Specific Aim 1: To examine the impact of a wawokiya health advocate (WHA) palliative care intervention on patient health outcomes including quality of life, symptom burden, and psychosocial wellbeing.

H1: Compared to patients in the waitlist group, patients enrolled in the WHA intervention will have a better quality of life, greater psychosocial wellbeing, and lower symptom burden.

Specific Aim 2: To assess the impact of a WHA palliative care intervention on patient healthcare utilization including emergency room visits, hospitalizations, telehealth visits, and concordance of services with goals of care.

H2: Patients enrolled in the WHA intervention will have fewer ER visits and hospitalizations and a greater number of telehealth visits than patients enrolled in the waitlist group.

H3: A greater proportion of patients enrolled in the WHA intervention will die in their preferred location.

Specific Aim 3: To examine the impact of a WHA palliative care intervention on caregiver outcomes including coping, caregiver burden, and quality of life.

H4: Compared to caregivers in the waitlist group, caregivers enrolled in the WHA intervention will have a better quality of life, better coping, and decreased caregiver burden.

Specific Aim 4: To explore moderators and mediators of a WHA as a palliative care navigator on rural reservations in South Dakota.

H5: Adherence to protocols will moderate the effectiveness of a WHA as a PC navigator.

.

DETAILED DESCRIPTION:
One of the greatest areas of need in cancer care for American Indians in the Northern Plains is palliative care.Defined as the services needed to live well with serious illness, access to palliative care services by this population is almost non-existent, particularly in areas like western South Dakota where many tribal lands are located. Because of the distance to the nearest cancer care facility, the lack of transportation, and the lack of community-based palliative care, the great majority of American Indians with cancer living on Reservations are separated from their families during inpatient cancer care and die either alone in a hospital or at home suffering unnecessarily from symptoms such as pain, shortness of breath and anxiety. While this would be unacceptable for any group, it is particularly detrimental for Tribal Nations in the Northern Plains given the US governmental responsibility for providing their health care, the poverty experienced by the tribes, and the importance the people of these Nations place on spiritual preparation and community support at the end of life.

The past decade has witnessed substantial advances in the delivery of palliative care in other settings, particularly urban areas. Early application of palliative care services has been demonstrated to improve outcomes for patients with cancer, and new models of palliative care delivery are being developed, tested and implemented. Key features of these models, including the use of primary palliative care education, patient navigators and telemedicine for palliative care, have clear applications in the delivery of palliative care to American Indians in the Northern Plains.

Over the last 7 years, investigators have developed a multidisciplinary, Native-driven collaboration to advance the health of Lakota tribes that brings together multiple organizations in South Dakota (Great Plains Tribal Leaders Health Board [GPTLHB], Avera Health, Walking Forward, South Dakota State University School of Nursing, Indian Health Service [IHS]), the three largest tribes in western South Dakota (Cheyenne River, Oglala, and Rosebud Sioux tribes) and Mass General/Harvard. Initially developed to support clinical care for the Rosebud Sioux tribe, the Great Plains Lakota Health Research Collaboration (GPLHRC) has expanded to address critical health care issues affecting tribal communities across the region.

In the initial phase of the current project, the GPLHRC engaged with community members from each of the three tribes to better understand the existing palliative care landscape. We held 19 talking circles with cancer patients and their caregivers and conducted 12 interviews with local tribal leaders and traditional healers. In addition, we interviewed 38 health care providers both on and off the reservations. In holding open discourse with these key stakeholders, the GPLHRC identified many of the needs and concerns held within the South Dakota provider and patient community regarding palliative care for reservation-dwelling individuals and several challenges providers and their patients face to accessing and/or delivering palliative care.

Our work revealed that the fragmentation of services between the IHS and the urban or semi-urban cancer centers, as well different cultural backgrounds of providers and American Indian patients significantly influence the delivery of palliative services. The need for better coordination between providers and improved navigation of palliative care resources for patients was highlighted across the community. Additionally, providers expressed a desire for additional knowledge about Lakota culture as well as additional knowledge about existing resources and health infrastructure on the reservations.

Informed by Community Advisory Board (CAB) and the qualitative data described above, the investigators have developed a wawokiya health advocate (WHA)-based palliative care navigation intervention that aims to improve the wellbeing of patients with cancer. After receiving a specialized training curriculum through the Harvard Medical School Center for Palliative Care (HMS CPC), WHAs will make regular home visits to patients suffering from cancer to assess needs and locate resources to appropriately address the issues assessed. In alignment with community feedback, patients and their caregivers will be allocated to a waitlist group or the intervention as dictated by WHA patient panel capacity. By evaluating the impact of the intervention on patients and caregivers compared to usual oncologic care, investigators aim to provide evidence for the long-term implementation of a sustainable approach to palliative care delivery for Reservation-dwelling American Indians in the Northern Plains and generate data to improve the quality of cancer care in rural settings across the US.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Age greater than or equal to 18 years old
* Carry an active invasive cancer diagnosis (other than non-melanoma skin cancer)
* Self-report as a member of a federally recognized tribe
* Reside on Pine Ridge, Rosebud, or Cheyenne River Indian Reservations or within the Contract Health Service Delivery Area of the Pine Ridge, Cheyenne River, or Rosebud IHS Service Unit
* Able to complete baseline surveys
* Able to provide informed consent
* A clinician responds "no" to the question: "Would it be a surprise if this person died in the next 12 months?"

Exclusion Criteria:

* Do not meet any of the above criteria

Caregivers

Inclusion Criteria:

* Are greater than or equal to 18 years old
* Reside in Pine Ridge, Rosebud, or Cheyenne River Indian Reservations or within the Contract Health Service Delivery Area of the Pine Ridge, Cheyenne River, or Rosebud IHS Service Unit
* Identified as caregiver by an enrolled patient;
* Caregiver will be defined as anyone who patients identify as a consistent source of physical, mental, emotional or spiritual support.
* Able to complete baseline survey
* Able to provide informed consent

Exclusion Criteria:

* Do not meet any of the criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cancer patient quality of life | Through study completion post baseline, an average of 1 year
  Change from baseline in patient-reported quality of life measured by the Functional Assessment of Cancer Therapy - General 7 (FACT-G7) through study completion (we anticipate an average of 1 year). FACT-G7 is a 7-item Likert scale (range 0-4). Scores range from 0-28, higher scores indicate better quality of life.
Cancer patient symptom burden | Through study completion post baseline, an average of 1 year
  Change from baseline in patient-reported symptom burden as measured by the Edmonton System Assessment System - revised (ESAS-r). The ESAS-r is a 9-item scale that measures a total of 9 symptoms on a continuous scale of 0 (no symptoms present) to 10 (most severe level). Scores range from 0-90. Higher scores indicated greater symptom burden.
Cancer patient loneliness | Through study completion, an average of 1 year
  Change from baseline in patient-reported loneliness as measured by the University of California-Los Angeles (UCLA) three-item loneliness scale. The UCLA loneliness scale is a 3-item likert scale (range 1-3). Scores range from 3-9. Higher scores indicate greater loneliness.
Cancer patient hope | Through study completion, an average of 1 year
  Change from baseline in patient-reported hope as measured by Herth Hope Index (HHI). The HHI is a 12-item Likert scale (1-4). Scores range from 12-28. Higher scores indicate higher levels of hope.

SECONDARY OUTCOMES:
Hospital Admissions | Through study completion, an average of 1 year
  Number of times patient is hospitalized overnight
ER Visits | Through study completion, an average of 1 year
  Number of separate trips to Emergency Room
Telemedicine VIsits | Through study completion, an average of 1 year
  Number of visits with a provider over video or phone call
Home Visits (not related to study) | Through study completion, an average of 1 year
  Number of home visits with a health care professional (not a wawokiya/study interventionist)
Caregiver Quality of life | Through study completion, an average of 1 year
  Change from baseline in caregiver-reported quality of life across 10 domains as measured by the CareGiver Oncology Quality of Life questionnaire (CarGOQOL). The CarGOQOL is a 29-item Likert scale (1-5). Scores range from 29- 145. Higher scores indicate a higher quality of life.
Caregiver burden | Through study completion, an average of 1 year
  Change from baseline in caregiver-reported burden measured by the Montgomery Borgatta Caregiving Burden (MBCB). The MBCB is a 14-item Likert scale (15) subdivided into 3 scales(objective burden, subjective stress burden, subjective demand burden). Scores on the objective subscale range from 6-30 and scores on the stress and demand burden subscales range from 4-20. Higher scores across sub scales indicate higher burden.
Caregiver loneliness | Through study completion, an average of 1 year
  Change from baseline in caregiver-reported loneliness as measured by the University of California-Los Angeles (UCLA) three-item loneliness scale. The UCLA loneliness scale is a 3-item Likert scale (range 1-3). Scores range from 3-9. Higher scores indicate greater loneliness.
Caregiver hope | Through study completion, an average of 1 year
  Change from baseline in caregiver-reported hope as measured by Herth Hope Index (HHI). he HHI is a 12-item Likert scale (1-4). Scores range from 12-28. Higher scores indicate higher levels of hope.

OTHER OUTCOMES:
WHA Intervention Fidelity | Through study completion, an average of 1 year
  Adherence to protocol will be evaluated via semi-structured interviews with patients

CONTACTS AND LOCATIONS:
Locations (1):
- Walking Forward - Avera Research Institute, Rapid City, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers who are not involved in this study.